CLINICAL TRIAL: NCT02836067
Title: Impact of Smoking and Its Cessation on Systemic and Airway Immune Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-35295; R01DA042685-02 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: HIV; Smoking
MeSH Terms: conditions — Smoking | interventions — Counseling; Bronchoscopy; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Smokers (Other): HIV-positive smokers will be enrolled in a smoking cessation program including the following procedures:
  Counseling Smoking cessation drugs Questionnaires Blood Draw Bronchoscopy
  Interventions: Behavioral: Counseling; Other: Smoking Cessation drugs; Procedure: Bronchoscopy; Procedure: Blood Draw; Behavioral: Questionnaires
- Non-Smokers (Other): HIV-positive non-smokers will be enrolled as a comparison group to HIV-positive smokers and will have the following procedures:
  Questionnaires Blood Draw Bronchoscopy
  Interventions: Procedure: Bronchoscopy; Procedure: Blood Draw; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Counseling — Smoking cessation counseling
  Arms: Smokers
Other: Smoking Cessation drugs — Medication to aid smoking cessation
  Arms: Smokers
Procedure: Bronchoscopy — Bronchoscopy
Procedure: Blood Draw — Screening and research blood draws
Behavioral: Questionnaires — Behavioral questionnaires

SUMMARY:
The purpose of this study is to learn how smoking affects the immune systems in people with HIV infection. The investigators would like to know if HIV infected smokers who quit smoking have different responses in their tissues from people who keep smoking.

DETAILED DESCRIPTION:
For Aim 1, a total of up to 30 patients with HIV disease who have never smoked will be recruited, with recruitment stopping before 30 samples if the samples from 20 patients that can be used in analysis have been obtained. These 20 non-smoker samples will be compared to those of 20 active smokers with HIV disease, without evidence of COPD from spirometry, who are matched in demographics. Smokers who are interested in participating in a smoking cessation program will be referred to our Clinical Trials Unit (CTU) for all subsequent study visits.

Additionally, a comparison group of 20 uninfected smokers who have already been enrolled in the co-investigator's (Dr. Kwon) study will be used as comparison group. These participants have similar inclusion/exclusion criteria as this study and have been verified to be HIV-antibody negative. The investigators will obtain de-identified samples and immunological and virological data already collected by Dr. Kwon. De-identified banked PBMC, plasma and BAL samples will also be accessible to us using a material transfer agreement to perform epithelial transcriptional gene expression profiling.

For Aim 2, a total of 100 HIV-infected individuals on effective ART who are active smokers and interested in participating in a smoking cessation program will be recruited. If 30 individuals who achieve 10-week of cessation are enrolled before 100 HIV smokers are fully enrolled, enrollment will cease, as 100 participants is an overestimate of the number of patients needed need to enroll to have 30 subjects achieve successful smoking cessation. Just like for nonsmokers, recruitment for both smoker cohorts will stop before 30 if samples from 20 patients that can be used in analysis have been obtained. The maximum total number of patients needed for the grant is 130 (100 HIV smokers, 30 HIV non-smokers).

About130 participants will be recruited from the BMC Center for Infectious Diseases (CID) outpatient clinic, other outpatient clinics within BMC, affiliated community health centers (CHCs), BWH, MGH, Tufts Medical Center, and Beth Israel Deaconess Medical Center. The BMC CID clinic serves the largest HIV-infected population in Boston, approximately 1,700 persons, and is composed largely of an urban socioeconomically disadvantaged population. Over 50% of HIV-infected patients in the CID are smokers, and >60% (based on prescription history of NRT, bupropion, varenicline) have attempted smoking cessation. Participants will be recruited from flyers, the BMC ReSPECT registry, medical record screening, and physician referrals.

ELIGIBILITY:
Inclusion criteria.

1. HIV infected on ART ≥ 6 months
2. Virologically suppressed (<50 cop/ml) at the time of enrollment (lab test within 3 months )
3. Smoking Status:

   Currently Active Smoker: Self-reported regular cigarette use with positive cotinine test at screening visit.

   OR Non-smoker: self-reported non-smokers confirmed by negative cotinine test at screening visit.
4. Laboratory values within 3 months prior to enrollment that meet the following criteria:

   1. Hemoglobin ≥ 8.0 g/dL
   2. Platelet count ≥ 80,000/mm3
5. For females of child-bearing potential: Negative urine pregnancy test (sensitive to 25 IU HCG) at screening visit.

For purposes of this study, a female is considered of child-bearing potential unless:

* Permanently sterile (includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy)
* Medically documented ovarian failure
* Post-menopausal, defined as ≥ 55 years of age with cessation of menses for ≥ 12 months

Exclusion criteria:

1. Pregnant or breast-feeding or less than 8 weeks post-partum.
2. Active malignancy and receiving concurrent treatment (i.e. chemotherapy, radiation therapy, investigational treatment).
3. Significant immunological illnesses/deficiencies
4. Recent active illness within the past 1 month (i.e. respiratory viral infection, pneumonia, bacterial infections, bone infection)
5. History of tuberculosis, lung cancer, bronchiectasis, pulmonary fibrosis, or pulmonary hypertension
6. Self-reported regular or recreational use of inhaled substances (such as marijuana, crack, fentanyl, heroin, hookah, e-cigarettes) as well as chewing tobacco within past month. Reports of no such use within the past month will be confirmed by a urine tox screen performed at the Screening Visit.
7. Self-reported regular use of inhaled substances (such as crack, fentanyl, heroin, hookah, e-cigarettes) in the past (prior to 1 month ago and within the past 5 years), with use occurring for > 1 year. (Marijuana use is allowable.)
8. Spirometry criteria FEV1/FVC < 0.7 (definition of COPD) and GOLD (severe-very severe) Stage 3 or 4 within past 12 months
9. A history of alcohol dependence within the 6 months prior to enrollment
10. History of intolerance, sensitivity, allergy or anaphylaxis to lidocaine or other amide anesthetics, as well as benzocaine or other ester type anesthetics
11. History of recent myocardial infarction (within past 6 months). Non-coronary ischemia MI is allowed (i.e. cocaine-induced)
12. Chronic renal failure requiring dialysis
13. Decompensated cirrhosis
14. Currently taking anticoagulants including but not limited to: heparin (Hep-Lock, Hep-Pak), Hep-Pak CVC, Heparin Lock Flush), warfarin (Coumadin), tinzaparin (Innohep), enoxaparin (Lovenox), danaparoid (Orgaran), dalteparin (Fragmin), clopidogrel (Plavix), prophylactic aspirin, and NSAID use and unable to stop for 48 hours prior to bronchoscopy
15. Taking any of the following medications within 30 days prior to enrollment: systemic steroids (inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (e.g., local injection of interferon alpha for treatment of HPV is permitted) or systemic chemotherapy, anti-TNF agents
16. Recent abdominal surgery (within past 3 months)
17. Recent eye surgery (within past 3 months)
18. Investigator discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
.Difference in T cell and monocyte immune subsets, level of activation | Week 12
  Aliquots of BAL and PBMC will be stained for surface antibodies to distinguish differentiation and activation markers. Monocyte cells will be phenotyped by CD3, CD19 and CD56 all on FITC, CD14 BUV 395, CD16 BV510, CCR2 PE, CX3CR1 APC, CD11c PEcf594, CD80 BV 421, CD86 BV 605, HLA-DR BV785, CD123 PE Cy7 and eFluor780 fixable viability dye. T cell populations will be stained for CD3, CD4, CD8, CD45RA, CCR7, CD27 and CD28; activation status by expression of CD25, CD38, CD69, HLA-DR, OX40. We will determine if they are Th2/Tc2-type cells by expression of CCR4, CCR8, T1/ST2, CRTH2. Flow will be performed on a LSRII (BD) and analyzed with FlowJo (Tree Star).

SECONDARY OUTCOMES:
Difference in levels of plasma inflammatory markers | Week 12
  For analysis of inflammatory protein levels, BAL fluid will be concentrated 10-fold using a Centricon filter (Millipore) with a 3,000 MW cutoff. We have found that assaying for cytokines is more reliable when the BAL is concentrated 10-fold since BAL is diluted ~100-fold by the procedure. sCD14 (R&D) and iFABP (Hycult) will be measured by ELISA. LPS will be measured with the LAL assay (Pierce) and sCD163 (Trillium Diag). Additional human cytokines associated with inflammatory processes, including TNF-α, IFN-α/g, IL-6/7/10, IP-10 and MCP-1, will be measured using the Milliplex cytokine- kit (Millipore), read on a Luminex 100 and analyzed with Beadview software (Upstate Cell).
Differences in level of oxidative stress | Week 12
  Cells from blood and BAL will be stimulated with and without PMA for 30 min. and incubated with DHR123 to directly detect intracellular ROS production. Cells will be stained with fluorescent antibodies recognizing lineage markers for T cells (CD3, CD4, CD8), macrophages (CD14), B cells (CD19, CD20), and granulocytes (CD66b).
Differences in the level of measure of HIV residual viremia | Week 12
  Measure levels of HIV-1 ca-DNA, ca-RNA and 2-LTR circles in BAL and PBMC samples collected from HIV-infected smokers versus non-smokers. Cellular DNA and RNA from PBMCs and BAL cells will be extracted with AllPrep DNA/RNA mini kit (Qiagen). HIV-1 ca-DNA will be quantified using a sensitive quantitative PCR (qPCR) assay to measure a conserved LTR/gag region96, and modified in our lab118. Measurements of ca-DNA will be reported as copies of HIV DNA/106 cells. Quantification of a conserved region of the human CCR5 will be used to determine the number of cells in each sample well.
Differences airway transcriptional profile | Week 12
  Compare gene expression profiles between HIV smokers and non-smokers. Library preparation for RNA sequencing will be accomplished using Illumina's TruSeq RNA Sample Prep Kit v2, using 200-500ng of total RNA from each bronchial epithelial brushing. Briefly, RNA will be isolated using poly(A) selection, fragmented into a range of lengths centered around 200 base pairs, and randomly primed for reverse transcription followed by first and second-strand synthesis to create double-stranded cDNA fragments. Subsequently, these fragments will undergo PCR amplification, purification, and be used for cluster generation on a cBot machine using Illumina TruSeq Paired-End Cluster Generation Kits.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Asundi, M.D., Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02836067/ICF_000.pdf